CLINICAL TRIAL: NCT00172354
Title: Hydrocortisone in Patients of Out-of-hospital Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 930502
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Heart Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is an important issue for the emergency physicians and co-workers. How to improve the return of spontaneous circulation (ROSC) rate and prognosis of these patients challenges the emergency team. When encounters stress, the hypothalamus of human releases corticotropin releasing hormone, which in turn stimulates the pituitary gland to release ACTH. Then ACTH acts on the adrenal gland to release glucocorticoid to against stress. Foley PJ et al found the dogs with bilateral adrenalectomy had lower ROSC rate during resuscitation than those without surgery[1]. Karl H. Linder et al showed OHCA patients had high serum vasopressin and ACTH level but low serum cortisol level. Besides, the serum cortisol level had a negative correlation with collapse duration (no CPR duration)[2]. Studies also revealed the successfully resuscitated patients had higher serum ACTH and cortisol level than non-resuscitated ones[2,3]. In addition, the serum cortisol level was found to be correlated with short term survival rate and hemodynamic status in resuscitated OHCA patients[3]. Animal study also showed mice receiving higher dosage of hydrocortisone had higher ROSC rate and lower epinephrine requirement than those receiving lower dosage of hydrocortisone or normal saline.

<Reference>

1. Foley PJ, Tacker WA, Wortsman J, Frank S, Cryer PE.;" Plasma catecholamine and serum cortisol responses to experimental cardiac arrest in dogs."Am J Physiol 1987;253:E283-9
2. Lindner KH, Strohmenger HU, Ensinger H, Hetzel WD, Ahnefeld FW, Georgieff M.;" Stress hormone response during and after cardiopulmonary resuscitation."Anesthesiology 1992;77:662-8
3. Schultz CH, Rivers EP, Feldkamp CS, Goad EG, Smithline HA, Martin GB, Fath JJ, Wortsman J, Nowak RM.;"A characterization of hypothalamic-pituitary-adrenal axis function during and after human cardiac arrest."Crit Care Med 1993;21:1339-47
4. Smithline H, Rivers E, Appleton T, Nowak R.;"Corticosteroid supplementation during cardiac arrest in rats."Resuscitation 1993;25:257-64

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest

Exclusion Criteria:

* pregnancy
* younger than 18 years old
* trauma
* concurrent steroid use
* ECMO use in resuscitation
* allergy to steroid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-10; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jone Chen, PhD, Study Director — Chiarman of NTUH emergency department
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan